CLINICAL TRIAL: NCT04283695
Title: A Phase 1, Open-labeled, Single-dose, One-sequence, One-period, 3-part Study to Investigate the Absorption, Metabolism, Excretion, Absolute Bioavailability, and Immunogenicity of GX-I7 in Healthy Volunteers
Brief Title: To Investigate the Absorption, Metabolism, Excretion, Absolute Bioavailability, and Immunogenicity of GX-I7 in Healthy Volunteers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Howard Lee, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Mab_GX_I7
Record Dates: First submitted 2019-11-18; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Leukopenia
MeSH Terms: conditions — Leukopenia | interventions — efineptakin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): IM: GX-I7 60 µg/kg IV: [14C]-GX-I7 40 µg
  Interventions: Drug: GX-I7 or [14C] GX-I7
- Part 2 (Experimental): IV: [14C]-GX-I7 40 µg
  Interventions: Drug: GX-I7 or [14C] GX-I7
- Part 3 (Experimental): IM: GX-I7 60 µg/kg, [14C]-GX-I7 40 µg
  Interventions: Drug: GX-I7 or [14C] GX-I7

INTERVENTIONS:
Drug: GX-I7 or [14C] GX-I7 — IM GX-I7 or IV/IM microdose of GX-I7

SUMMARY:
A Phase 1, open-labeled, single-dose, one-sequence, one-period, 3-part study to investigate the absorption, metabolism, excretion, absolute bioavailability, and immunogenicity of GX-I7 in healthy volunteers

DETAILED DESCRIPTION:
A Phase 1, open-labeled, single-dose, one-sequence, one-period, 3-part study to investigate the absorption, metabolism, excretion, absolute bioavailability, and immunogenicity of GX-I7 in healthy volunteers To show ABA and Mass balance of GX-I7

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to give informed consent after listening character of the clinical trial
2. Must be 19-45 years of age, inclusive
3. Weight 50-100kg, BMI 18-30kg/m2
4. Subject who is adequately able to attend the study based on medical history and physical exam, no clinically significant abnormality from vital sign and clinical laboratory values
5. No clinical abnormality from ECG test
6. Non-smoker (no smoking or no use of any product containing nicotine least for one month and negative from urine test)

Exclusion Criteria:

1. Suspected or confirmed malignancy, or has malignancy history
2. Any clinically significant acute or chronic medical condition requiring care of a physician, in liver, biliary tract, renal, nervous system (CNS or peripheral). respiratory system, endocrine (diabetes, hyperlipidemia etc), cardiovascular (congestive heart failure, coronary artery disease, myocardial infarction etc), hematology, malignancy, urinary disease, mental disorder, musculoskeletal disorder, immune system (rheumatoid arthritis, lupus etc), otorhinolaryngologic diseases
3. Positive to HBsAg, hepatitis C virus (HCV) Ab and HIV Ab
4. Are considering or scheduled to undergo any surgical or dental procedure during the study
5. Administered other Investigational Product (IP) by attending other clinical study or biological equivalent study within recent 6 months
6. Any Serious adverse drug reaction (SAR) against vaccines or antibiotics, any medical history with serious allergic diseases
7. Positive from urine drug screen or respiratory alcohol screen at medical screening
8. History of alcohol, drug, or substance abuse in the past 12 months
9. A heavy alchol consumer (>21 units/week, 1 unit = 10 g of pure alcohol) or Consumption of alcohol within 48 hours prior to hospitalization
10. Medications with antacid, analgesic, herbal treatment, vitamin, mineral (except maximum 4 grams of acetaminophen) hormone, steroids, insulin, hypoglycemic drug or other hormone substitute within 14 days before administration
11. Planning pregnancy or donation of sperm/disagreeing proper contraception during the study and 3 months following IP administration
12. Do not have veins suitable for cannulation or multiple venipunctures
13. Previously donate whole blood within 60 days or component blood within 14 days
14. Excessive consumption of foods containing grapefruits
15. Any other factor that the Investigator thinks will increase subject risk with participation

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Total radioactivity at feces,urine,blood to measure total recovery rate | 29 days
  radioactivity in nCi

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea